CLINICAL TRIAL: NCT05390151
Title: LATFIA-trial: Laser Assisted Treatment of Fistula In Ano Randomized Controlled Trial Comparing FiLaCTM to Rectal Advancement Flap
Brief Title: Laser Assisted Treatment of Fistula In Ano
Acronym: LATFIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universitair Ziekenhuis Brussel (Other); University Hospital, Ghent (Other); AZ St.-Dimpna Geel (Other); Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 000202
Record Dates: First submitted 2022-04-21; First posted 2022-05-25 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-03

CONDITIONS: Fistula in Ano; Rectal Fistula
Keywords: Rectal, Advancement Flap; Laser assisted Fistula Closure; Randomised Control Trial
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser assisted fistula closure (Active Comparator): Group to be actively treated with laser assisted fistula surgery
  Interventions: Procedure: Laser treatment of anal fistula
- Rectal advancement flap (Active Comparator): Group to be actively treated with a rectal advancement flap.
  Interventions: Procedure: RAF

INTERVENTIONS:
Procedure: Laser treatment of anal fistula — using a radial laserprobe to treat transsphincteric fistula
  Other Names: FiLAC - LAFT
  Arms: Laser assisted fistula closure
Procedure: RAF — current golden standard in transsphincteric fistula surgery
  Other Names: rectal advancement flap
  Arms: Rectal advancement flap

SUMMARY:
Randomised Controlled Trial comparing Laser assisted closure of transsphincteric fistula to the rectal advancement flap.

DETAILED DESCRIPTION:
A prevalent and complex fistula type is the high transsphincteric (TS) fistula. It typically runs through the upper two-thirds of the external anal sphincter (EAS) and is, due to the high risk of fecal incontinence, not suitable for fistulotomy and sphincter sparing treatment is required. To be included in this trial the participants should have a single, continuous TS fistula of cryptoglandular origin, that is treated by loose seton drainage for at least 2 months and is mapped by MRI. Participants with IBD, hidradenitis suppurativa or a malignant fistula will be excluded. Intervention Fistula Laser Closing (FiLaCTM) (Biolitec, Germany) is an endofistular technique, using a radial-emitting laser fiber that emits laser light with a maximum penetration depth of 2 - 3 mm. It destroys both the crypt gland and the additional epithelial layer of the fistula without damaging the sphincter. The fiber is inserted until the internal opening, activated and pulled backwards slowly, allowing the laser to have its effect. The external opening is excised and the internal opening is closed with a single absorbable suture. Rectal advancement flap is currently the gold standard for sphincter sparing treatment of high transsphincteric fistulae. The fistula is cored out and an advancement flap is made of mucosa and submucosa. The opening of the fistula in the flap is excised, the residual internal opening is closed with absorbable suture and the flap is sutured below the fistula to the anoderm. The advancement flap is a difficult technique that requires a relatively large transanal dissection that results in postoperative pain and may lead to disturbances in continence. Preliminary results with the Filac technique show fistula healing rates comparable to the advancement flap. Due to its simplicity, speed and minimal invasiveness the investigators expect a benefit for the participants in terms of postoperative pain, operating time and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with fistula involving more than one-third of the external anal sphincter
* Single, continuous fistula tract at time of inclusion
* Loose seton present in fistula tract for 2 months or more at time of inclusion
* Age ≥ 18
* Able to complete an informed written consent, understand its implications and contents, and participate in follow-up

Exclusion Criteria:

* Fistula tract < 1 cm
* Complex fistula tract system (branching of fistula tract inside the sphincter complex)
* Pregnancy
* HIV-positive
* Crohn´s disease, Ulcerative colitis
* Fistula due to malignancy
* Tuberculosis
* Hidradenitis Suppurativa
* No internal opening
* Unable to undergo or contraindications to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Primary fistula closure after index laser or flap treatment | 6 months
  Success rate (number of patients) of laser/flap treatment defined as full healing (fistula closure) after the index procedure

SECONDARY OUTCOMES:
Secondary Fistula closure | 6 months
  Secondary success rate (number of patients) defined as full healing (fistula closure) after a second procedure (either rectal advancement flap, laser treatment, fistulotomy)
Postoperative Pain | 6 months
  Reported pain after laser or flap treatment: measured using the visual analog scale - VAS where 0 = no pain; 10 = worst pain imaginable,
Postoperative fecal incontinence | 6 months
  Reported fecal incontinence after laser or flap treatment:
  measured using the Vaizey score where minimum score 0 = perfect continence; maximum score 24 = totally incontinent)
Postoperative wound complications | 6 months
  Reported wound complications after laser or flap treatment defined as wound dehiscence or bleeding as reported on the adverse event forms
Postoperative Quality of Life | 6 months
  General postoperative well being and ability to partake in daily life and daily tasks (specific role functioning) measured and scored using the SF 36 questionnaire (consisting of 8 weighted scales:
  vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role, functioning, and mental health. The lower the score the more disability. The higher the score the less disability)
  This outcome is measured in all participants after the initial procedure (index flap or laser treatment) as well as after a second procedure (in case of recurrence)
Primary Recurrence | 6 months
  Number of participants presenting with a clinical recurrence or residual fistula after initial and laser/flap treatment (index procedure)
Secondary Recurrence | 12 months
  Number of participants presenting with a clinical recurrence or residual fistula after the second procedure (Laser - Flap - Fistulotomy - Ligation of the fistula tract, video-assisted fistula treatment)
Identify predictive factors for clinical fistula healing to determine the treatment indications. | 6 months
  This outcome evaluates the correlations between patients'/ fistula's clinical characteristics and primary healing rates

CONTACTS AND LOCATIONS:
Overall Officials: Niels Komen, M.D. Phd, Study Chair — University Hospital, Antwerp; Sander Van Hoof, M.D., Principal Investigator — University Hospital, Antwerp
Locations (5):
- Belgium (5):
  - Antwerp University Hospital, Edegem, Antwerpen
  - Az St Dimpna Geel, Geel, Antwerpen
  - Jessa Ziekenhuis Hasselt, Hasselt, Limburg
  - Gent University Hospital, Ghent, Oost- Vlaanderen
  - Brussels University Hospital, Brussels

IPD SHARING:
Plan to Share IPD: No